CLINICAL TRIAL: NCT05610514
Title: Pulmonary and Cardiac Effects of E-Cigarette Use in Pulmonary Patients Who Smoke Cigarettes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Diann Gaalema, Associate Professor, Department of Psychiatry, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000511; U54DA036114-07 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Asthma-COPD Overlap Syndrome
Keywords: chronic obstructive pulmonary disease; pulmonary; cardiac; cigarettes; e-cigarettes; smokers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema; Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combustible Cigarette (No Intervention): Participants in this arm will smoke their usual brand of combustible cigarettes for two weeks.
- E-Cigarette (Experimental): Participants in this arm will smoke electronic cigarettes for two weeks. E-cigarettes (either JUUL or Vuse Alto) and pods (JUUL: Virginia tobacco flavor at 3% or 5% nicotine concentration; Vuse Alto: golden tobacco flavor at 1.8%, 2.4%, or 5% nicotine concentration) will be provided.
  Interventions: Other: E-Cigarette; Behavioral: Financial Incentives

INTERVENTIONS:
Other: E-Cigarette — Altering the availability of e-cigarettes
  Arms: E-Cigarette
Behavioral: Financial Incentives — Altering the availability of financial incentives for abstaining from combustible cigarettes
  Arms: E-Cigarette

SUMMARY:
The purpose of this study is to compare the effects of e-cigarettes and continued smoking on pulmonary and cardiac outcomes in a population with established pulmonary disease.

DETAILED DESCRIPTION:
E-cigarettes with nicotine can affect important cardiopulmonary outcomes and likely pose less risk than cigarettes, but they are not harmless. Given the existing literature, there is a need for controlled trials of e-cigarette use in populations with cardiopulmonary disease to fill the gaps between these existing examinations. Clarifying how the pulmonary and cardiac effects of e-cigarettes compare to use of conventional cigarettes in those with cardiopulmonary disease beyond single acute exposures will provide important new health information that can help inform policy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40 years of age or older
* Current, every day smoker (5 or more cigarettes per day for one year or longer) confirmed with intake CO of 8ppm or greater
* Established pulmonary disease (chronic obstructive pulmonary disease [COPD], chronic bronchitis, emphysema, or asthma-COPD overlap syndrome) confirmed by physician diagnosis and/or current prescription of medication for treatment (i.e., LABA, LAMA, +/- ICS, or combination)
* Lives and plans to remain in the greater Burlington, VT area for the next month
* No intention to quit smoking within the next month
* Speaks English

Exclusion Criteria:

* Patients who are medically unstable (unstable symptoms, changes in medications or hospitalizations within last 3 months)
* Inability to conduct in-home measurements.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Baseline FEV1/FVC Ratio | Intake assessment
  Ratio of the amount of air forced from the lungs in one second (Forced Expiratory Volume in the First Second; FEV1) to the amount of air forced from the lungs throughout an entire measurement (Forced Vital Capacity; FVC), as assessed via spirometry
Change from Baseline FEV1/FVC Ratio each day | Daily through study completion, an average of 4 weeks
  Ratio of the amount of air forced from the lungs in one second (Forced Expiratory Volume in the First Second; FEV1) to the amount of air forced from the lungs throughout an entire measurement (Forced Vital Capacity; FVC), as assessed via spirometry
Change from Baseline FEV1/FVC Ratio at 2 weeks | Assessment completed 2 weeks after intake assessment
  Ratio of the amount of air forced from the lungs in one second (Forced Expiratory Volume in the First Second; FEV1) to the amount of air forced from the lungs throughout an entire measurement (Forced Vital Capacity; FVC), as assessed via spirometry
Change from Baseline FEV1/FVC Ratio at 4 weeks | Assessment completed 4 weeks after intake assessment
  Ratio of the amount of air forced from the lungs in one second (Forced Expiratory Volume in the First Second; FEV1) to the amount of air forced from the lungs throughout an entire measurement (Forced Vital Capacity; FVC), as assessed via spirometry
Baseline Lung Reactance at 5Hz (X5) | Intake assessment
  Measurement of the ability of the lung to store energy, as measured by oscillometry
Change from Baseline Lung Reactance at 5Hz (X5) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Measurement of the ability of the lung to store energy, as measured by oscillometry
Change from Baseline Lung Reactance at 5Hz (X5) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Measurement of the ability of the lung to store energy, as measured by oscillometry
Baseline Lung Resistance at 5Hz and 19Hz (R5 and R19) | Intake assessment
  Airway impedence in the lungs as measured by oscillometry
Change from Baseline Lung Resistance at 5Hz and 19Hz (R5 and R19) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Airway impedence in the lungs as measured by oscillometry
Change from Baseline Lung Resistance at 5Hz and 19Hz (R5 and R19) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Airway impedence in the lungs as measured by oscillometry
Baseline Oxygen Saturation (SpO2) | Intake assessment
  Amount of oxygen carried in the blood as a percentage of the normal maximum, as assessed via pulse oximetry
Change from Baseline Oxygen Saturation (SpO2) each day | Daily through study completion, an average of 4 weeks
  Amount of oxygen carried in the blood as a percentage of the normal maximum, as assessed via pulse oximetry
Change from Baseline Oxygen Saturation (SpO2) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Amount of oxygen carried in the blood as a percentage of the normal maximum, as assessed via pulse oximetry
Change from Baseline Oxygen Saturation (SpO2) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Amount of oxygen carried in the blood as a percentage of the normal maximum, as assessed via pulse oximetry
Baseline Fractional Exhaled Nitric Oxide (FeNO) | Intake assessment
  Amount of nitric oxide in the breath
Change From Baseline Fractional Exhaled Nitric Oxide (FeNO) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Amount of nitric oxide in the breath
Change From Baseline Fractional Exhaled Nitric Oxide (FeNO) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Amount of nitric oxide in the breath
Baseline COPD Assessment Test Score | Intake assessment
  Score measuring the impact of COPD on an individual's life; scale of 0-40; higher score indicates worse outcome
Change from Baseline COPD Assessment Test Score at 2 weeks | Assessment completed 2 weeks after intake assessment
  Score measuring the impact of COPD on an individual's life; scale of 0-40; higher score indicates worse outcome
Change from Baseline COPD Assessment Test Score at 4 weeks | Assessment completed 4 weeks after intake assessment
  Score measuring the impact of COPD on an individual's life; scale of 0-40; higher score indicates worse outcome
Baseline St. George's Respiratory Questionnaire for COPD Patients Score | Intake assessment
  Score measuring the impact of COPD on overall health, daily life, and perceived well-being; scale of 0-100; higher scores indicate more limitations on overall health
Change from Baseline St. George's Respiratory Questionnaire for COPD Patients Score at 2 weeks | Assessment completed 2 weeks after intake assessment
  Score measuring the impact of COPD on overall health, daily life, and perceived well-being; scale of 0-100; higher scores indicate more limitations on overall health
Change from Baseline St. George's Respiratory Questionnaire for COPD Patients Score at 4 weeks | Assessment completed 4 weeks after intake assessment
  Score measuring the impact of COPD on overall health, daily life, and perceived well-being; scale of 0-100; higher scores indicate more limitations on overall health

SECONDARY OUTCOMES:
Baseline Blood Pressure | Intake assessment
  Force exerted by blood against the walls of the arteries
Change from Baseline Blood Pressure each day | Daily through study completion, an average of 4 weeks
  Force exerted by blood against the walls of the arteries
Change from Baseline Blood Pressure at 2 weeks | Assessment completed 2 weeks after intake assessment
  Force exerted by blood against the walls of the arteries
Change from Baseline Blood Pressure at 4 weeks | Assessment completed 4 weeks after intake assessment
  Force exerted by blood against the walls of the arteries
Baseline Heart Rate | Intake assessment
  Number of time the heart beats per minute
Change from Baseline Heart Rate each day | Daily through study completion, an average of 4 weeks
  Number of time the heart beats per minute
Change From Baseline Heart Rate at 2 weeks | Assessment completed 2 weeks after intake assessment
  Number of time the heart beats per minute
Change From Baseline Heart Rate at 4 weeks | Assessment completed 4 weeks after intake assessment
  Number of time the heart beats per minute

OTHER OUTCOMES:
Baseline Carbon Monoxide (CO) | Intake assessment
  Amount of carbon monoxide in the breath
Change from Baseline Carbon Monoxide (CO) each day | Daily through study completion, an average of 4 weeks
  Amount of carbon monoxide in the breath
Change from Baseline Carbon Monoxide (CO) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Amount of carbon monoxide in the breath
Change from Baseline Carbon Monoxide (CO) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Amount of carbon monoxide in the breath
Baseline Tobacco Use Questionnaire | Intake assessment
  Assess tobacco use history
Baseline Fagerstrom Test of Nicotine Dependence (FTND) | Intake assessment
  Survey assessing addiction to nicotine
Baseline Wisconsin Inventory of Smoking Dependence Motives - Brief (WISDM-Brief) | Intake assessment
  Survey assessing smoking dependence
Baseline Minnesota Tobacco Withdrawal Scale (MNWS) | Intake assessment
  Evaluates effects of smoking cessation; scale of 0-60; higher scores are a worse outcome
Change from Baseline Minnesota Tobacco Withdrawal Scale (MNWS) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Evaluates effects of smoking cessation; scale of 0-60; higher scores are a worse outcome
Change from Baseline Minnesota Tobacco Withdrawal Scale (MNWS) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Evaluates effects of smoking cessation; scale of 0-60; higher scores are a worse outcome
Baseline Questionnaire on Smoking Urges-Brief (QSU-Brief) | Intake assessment
  Assesses smoking urges; scale of 10-70; higher scores indicate greater urge to smoke
Change from Baseline Questionnaire on Smoking Urges-Brief (QSU-Brief) at 2 weeks | Assessment completed 2 weeks after intake assessment
  Assesses smoking urges; scale of 10-70; higher scores indicate greater urge to smoke
Change from Baseline Questionnaire on Smoking Urges-Brief (QSU-Brief) at 4 weeks | Assessment completed 4 weeks after intake assessment
  Assesses smoking urges; scale of 10-70; higher scores indicate greater urge to smoke
Daily Tobacco Use Questionnaire | Daily during each two-week arm of the study
  Measure tobacco use (cigarettes, e-cigarettes, smokeless tobacco) on a daily basis;
Health Changes Questionnaire at 2 week assessment | Assessment completed 2 weeks after intake assessment
  Assesses how health has changed since previous visit; 4 yes/no questions about whether there have been any changes in physical/mental health, changes in medications, access to medical care, or changes in normal routine in the last 24 hours; 1 question rating overall health on a scale of 1 to 10 with 10 being the best
Health Changes Questionnaire at 4 week assessment | Assessment completed 4 weeks after intake assessment
  Assesses how health has changed since previous visit; 4 yes/no questions about whether there have been any changes in physical/mental health, changes in medications, access to medical care, or changes in normal routine in the last 24 hours; 1 question rating overall health on a scale of 1 to 10 with 10 being the best

CONTACTS AND LOCATIONS:
Overall Officials: Diann E Gaalema, PhD, Principal Investigator — University of Vermont
Locations (1):
- Vermont Center on Behavior and Health, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No